CLINICAL TRIAL: NCT04332900
Title: Comparison of Immediate Effects of a Proximal and Distal Therapeutic Approach in Pain and Lower Limb Kinematic During Functional Tasks in People With Patellofemoral Osteoarthritis: A Crossover Study
Brief Title: Proximal and Distal Therapeutic Approach in Pain and Lower Limb Kinematic in People With Patellofemoral Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Larissa Rodrigues Souto, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2020/01599-7
Record Dates: First submitted 2020-02-16; First posted 2020-04-03 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Patellofemoral Osteoarthritis
Keywords: Knee osteoarthritis; Patellofemoral joint; Gait; Pain; Quality of life; Physiotherapy
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Foot Orthoses

STUDY DESIGN:
Intervention Model Description: randomised cross-over desing
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study only the person that will process and analyze the data could be blinded regarding the procedures and interventions of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control condition (No Intervention): In this condition there will not be any application of therapeutic approach.
- Intervention proximal condition (Experimental): The proximal therapeutic approach will be the SERF strap (S.E.R.F. strap; DonJoy Orthopedics, Inc., vista, CA).
  Interventions: Device: Elastic hip strap
- Intervention distal condition (Experimental): The distal therapeutic approach will be a pair of foot orthoses with semi-rigid arch support and medial elevation at the forefoot and at the rearfoot by 7° each (Propulsão Produtos Biomecânicos, Minas Gerais, Brazil).
  Interventions: Device: Insole

INTERVENTIONS:
Device: Elastic hip strap — The SERF Strap consist of a thin, elastic material that is secured to the proximal aspect of the leg, wraps in a spiral fashion around the thigh, and is anchored around the pelvis. The line of action of the SERF Strap pulls the hip into abdcution and external rotation.
  Other Names: S.E.R.F. Strap; DonJoy Orthopedics, Inc, vista, CA
  Arms: Intervention proximal condition
Device: Insole — Foot orthoses with semi-rigid arch support and medial elevation at the forefoot and at the rearfoot by 7° each that is made from a block of ethyl vinyl acetate with a thermo-moldable polymer (shore hardness of 45 A) and is manufactured through an automated computer numeric control machine (CNC routers).
  Other Names: Propulsão Produtos Biomecânicos, Minas Gerais, Brasil
  Arms: Intervention distal condition

SUMMARY:
This is a crossover study that will investigate the immediate effects of a proximal therapeutic approach (SERF strap) and a distal one (foot orthoses) on knee pain intensity, global change, symptoms, ease of performance and confidence after each task and lower limb kinematics (hip adduction and internal hip rotation peak, rearfoor eversion peak) during functional taks (level-ground walking and stepping manoeuvres) in people with patellofemoral ostheoartritis

DETAILED DESCRIPTION:
It will be enroled in this study 30 participants with patellofemoral ostheoartritis. The participants will be assessed during level walking at a self-selected speed and the stepping manoeuvre test under the three conditions that will be randomized: i) the control condition; ii) intervention proximal condition; and iii) intervention distal condition. The control condition refers to the condition in which no interventions will be administered. In both the intervention proximal condition and intervention distal condition, the respective therapeutic approach will be administered. For each functional task, three valid attempts will be collected. The primary outcome of this study is knee pain intensity and the secondary outcomes are both self-reported measures and kinematic variables measures. The self-reported measures are global change, symptoms, ease of performance and confidence, while the kinematic variables measures are hip adduction and internal hip rotation peak and rearfoor eversion peak

ELIGIBILITY:
Inclusion Criteria:

* Present anterior or retro patellar pain aggravated by two or more activities that overload the patellofemoral joint, such as going up and down stairs, squatting, remaining in the sitting position for long periods, getting up from the sitting position, kneeling or during physical exercise;
* Reporting pain of at least 3 on an 11-point scale (0 for no pain and 10 for the worst possible pain) during the activities described above and on most days during the last month;
* Have evidence of osteophyte formation in the patellofemoral joint on radiographs in the profile and axial skyline views through the Kellgren-Lawrence (K-L) grade ≥ 2, with minimal impairment in the tibiofemoral joint (KL <2);
* Body mass index (BMI) <35 Kg / m². Participants with unilateral or bilateral symptoms will be included in the study.

Exclusion Criteria:

* Current use or in the last 12 months of foot orthoses;
* Previous history of fracture or recurrent subluxation of the patella;
* Arthroscopic surgery or knee infiltrations in the last 3 months;
* Osteoarthritis known in other weight-bearing joints, including the spine;
* History of surgery on the hip, knee, ankle and foot joints;
* History of ankle sprain in the last 12 months;
* Osteotomy in the lower limbs;
* Current physical therapy in the lower limbs or in the last 6 weeks;
* Use of a cane or other walking aid;
* Any physical disability that is a contraindication for carrying out the evaluations and;
* Punctuation that suggests dementia according to the Mini-Mental State Examination, taking into account the education of the participants.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | The Pain intensity will be assessed immediately after the first valid attempt of the level-walking task in the Control Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the second valid attempt of the level-walking task in the Control Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the third valid attempt of the level-walking task in the Control Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the first valid attempt of the level-walking task in the Intervention Proximal Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the second valid attempt of the level-walkingtask in the Intervention Proximal Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the third valid attempt of the level-walking task in the Intervention Proximal Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the first valid attempt of the level-walking task in the Intervention Distal Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the second valid attempt of the level-walking task in the Intervention Distal Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the third valid attempt of the level-walking task in the Intervention Distal Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the first valid attempt of the stepping manoeuvre in the Control Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the second valid attempt of the stepping manoeuvre in the Control Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the third valid attempt of the stepping manoeuvre in the Control Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the first valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the second valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the third valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the first valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the second valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable
Pain intensity | The Pain intensity will be assessed immediately after the third valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  This variable will be collected using a visual analogue scale graduated in 100 millimeters, where the left end (zero) means no pain and the right end (ten) means the worst pain imaginable

SECONDARY OUTCOMES:
A global rating of change change (GRC) questionnaire | The GRC will be assessed immediately after the third valid attempt of the level-walking task in the Intervention Proximal Condition
  The GRC questionnaire is a 15 point self-report scale with criteria ranging from a 'very great deal worse' to a 'very great deal better.' The GRC is a valid and useful method for assessing the overall change in the quality of life of a person.
A global rating of change change (GRC) questionnaire | The GRC will be assessed immediately after the third valid attempt of the level-walking task in the Intervention Distal Condition
  The GRC questionnaire is a 15 point self-report scale with criteria ranging from a 'very great deal worse' to a 'very great deal better.' The GRC is a valid and useful method for assessing the overall change in the quality of life of a person.
A global rating of change change (GRC) questionnaire | The GRC will be assessed immediately after the third valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  The GRC questionnaire is a 15 point self-report scale with criteria ranging from a 'very great deal worse' to a 'very great deal better.' The GRC is a valid and useful method for assessing the overall change in the quality of life of a person.
A global rating of change change (GRC) questionnaire | The GRC will be assessed immediately after the third valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  The GRC questionnaire is a 15 point self-report scale with criteria ranging from a 'very great deal worse' to a 'very great deal better.' The GRC is a valid and useful method for assessing the overall change in the quality of life of a person.
Acceptable state of the patient's symptoms | The Acceptable state of the patient's symptoms will be assessed immediately after the third valid attempt of the level-walking tasks in the Intervention Proximal Condition
  The participants will answered this following question: "Considering your usual level of pain and also your functional impairment to perform tasks on a day-to-day basis, if you performed this functional task (gait or step-down test) with the application of this intervention (elastic band on the hip or foot orthosis) going forward, would you consider your current state to be satisfactory? " Participants will could answered "yes" or "no".
Acceptable state of the patient's symptoms | The Acceptable state of the patient's symptoms will be assessed immediately after the third valid attempt of the level-walking tasks in the Intervention Distal Condition
  The participants will answered this following question: "Considering your usual level of pain and also your functional impairment to perform tasks on a day-to-day basis, if you performed this functional task (gait or step-down test) with the application of this intervention (elastic band on the hip or foot orthosis) going forward, would you consider your current state to be satisfactory? " Participants will could answered "yes" or "no".
Acceptable state of the patient's symptoms | The Acceptable state of the patient's symptoms will be assessed immediately after the third valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  The participants will answered this following question: "Considering your usual level of pain and also your functional impairment to perform tasks on a day-to-day basis, if you performed this functional task (gait or step-down test) with the application of this intervention (elastic band on the hip or foot orthosis) going forward, would you consider your current state to be satisfactory? " Participants will could answered "yes" or "no".
Acceptable state of the patient's symptoms | The Acceptable state of the patient's symptoms will be assessed immediately after the third valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  The participants will answered this following question: "Considering your usual level of pain and also your functional impairment to perform tasks on a day-to-day basis, if you performed this functional task (gait or step-down test) with the application of this intervention (elastic band on the hip or foot orthosis) going forward, would you consider your current state to be satisfactory? " Participants will could answered "yes" or "no".
Ease of performing a task | The Ease of performing a task will be assessed immediately after the third valid attempt of the level-walking task in the Control Condition
  Participants will answer the following question: "How easy was this task?" and then they will respond according to the scale (markedly difficult; somewhat difficult; neither difficult nor easy; somewhat easy; markedly easy)
Ease of performing a task | The Ease of performing a task will be assessed immediately after the third valid attempt of the level-walking task in the Intervention Proximal Condition
  Participants will answer the following question: "How easy was this task?" and then they will respond according to the scale (markedly difficult; somewhat difficult; neither difficult nor easy; somewhat easy; markedly easy)
Ease of performing a task | The Ease of performing a task will be assessed immediately after the third valid attempt of the level-walking task in the Intervention Distal Condition
  Participants will answer the following question: "How easy was this task?" and then they will respond according to the scale (markedly difficult; somewhat difficult; neither difficult nor easy; somewhat easy; markedly easy)
Ease of performing a task | The Ease of performing a task will be assessed immediately after the third valid attempt of the stepping manoeuvre in the Control Condition
  Participants will answer the following question: "How easy was this task?" and then they will respond according to the scale (markedly difficult; somewhat difficult; neither difficult nor easy; somewhat easy; markedly easy)
Ease of performing a task | The Ease of performing a task will be assessed immediately after the third valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  Participants will answer the following question: "How easy was this task?" and then they will respond according to the scale (markedly difficult; somewhat difficult; neither difficult nor easy; somewhat easy; markedly easy)
Ease of performing a task | The Ease of performing a task will be assessed immediately after the third valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  Participants will answer the following question: "How easy was this task?" and then they will respond according to the scale (markedly difficult; somewhat difficult; neither difficult nor easy; somewhat easy; markedly easy)
Knee confidence | The knee confidence will be assessed immediately after the third valid attempt of the level-walking task in the Control Condition
  The knee confidence using a 100mm VAS, with the question phrased as "how confident did you feel completing that task? (terminal descriptors 0mm=very confident, 100mm=not confidente at all).
Knee confidence | The knee confidence will be assessed immediately after the third valid attempt of the level-walking task in the Intervention Proximal Condition
  The knee confidence using a 100mm VAS, with the question phrased as "how confident did you feel completing that task? (terminal descriptors 0mm=very confident, 100mm=not confidente at all).
Knee confidence | The knee confidence will be assessed immediately after the third valid attempt of the level-walking task in the Intervention Distal Condition
  The knee confidence using a 100mm VAS, with the question phrased as "how confident did you feel completing that task? (terminal descriptors 0mm=very confident, 100mm=not confidente at all).
Knee confidence | The knee confidence will assessed immediately after the third valid attempt of the stepping manoeuvre in the Control Condition
  The knee confidence using a 100mm VAS, with the question phrased as "how confident did you feel completing that task? (terminal descriptors 0mm=very confident, 100mm=not confidente at all).
Knee confidence | The knee confidence will be assessed immediately after the third valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  The knee confidence using a 100mm VAS, with the question phrased as "how confident did you feel completing that task? (terminal descriptors 0mm=very confident, 100mm=not confidente at all).
Knee confidence | The knee confidence will be assessed immediately after the third valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  The knee confidence using a 100mm VAS, with the question phrased as "how confident did you feel completing that task? (terminal descriptors 0mm=very confident, 100mm=not confidente at all).
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the stance phase of the level-walking of the first valid attempt in the Control Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the stance phase of the gait of the second valid attempt in the Control Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the stance phase of the level-walking of the third valid attempt in the Control Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the stance phase of the level-walking of the first valid attempt in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the stance phase of the level-walking of the second valid attempt in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the stance phase of the level-walking of the third valid attempt in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the stance phase of the level-walking of the first valid attempt in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the stance phase of the level-walking of the second valid attempt in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the stance phase of the level-walking of the third valid attempt in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the stance phase of the level-walking of the first valid attempt in the Control Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the stance phase of the level-walking of the second valid attempt in the Control Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the stance phase of the level-walking of the third valid attempt in the Control Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the stance phase of the level-walking of the first valid attempt in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the stance phase of the level-walking of the second valid attempt in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the stance phase of the level-walking of the third valid attempt in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the stance phase of the level-walking of the first valid attempt in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the stance phase of the level-walking of the second valid attempt in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the stance phase of the level-walking of the third valid attempt in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the stance phase of the level-walking of the first valid attempt in the Control Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the stance phase of the level-walking of the second valid attempt in the Control Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the stance phase of the level-walking of the third valid attempt in the Control Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the stance phase of the level-walking of the first valid attempt in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the stance phase of the level-walking of the second valid attempt in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the stance phase of the level-walking of the third valid attempt in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the stance phase of the level-walking of the first valid attempt in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the stance phase of the level-walking of the second valid attempt in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot of Eversion will be assessed during the stance phase of the level-walking of the third valid attempt in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the level-walking, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the first valid attempt of the stepping manoeuvre in the Control Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the second valid attempt of the stepping manoeuvre in the Control Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the third valid attempt of the stepping manoeuvre in the Control Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the first valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the second valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the third valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the first valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the second valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Adduction | The Lower limb kinematics - Peak of Hip Adduction will be assessed during the third valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the first valid attempt of the stepping manoeuvre in the Control Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the second valid attempt of the stepping manoeuvre in the Control Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the third valid attempt of the stepping manoeuvre in the Control Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the first valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the second valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the third valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the first valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the second valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Hip Medial Rotation | The Lower limb kinematics - Peak of Hip Medial Rotation will be assessed during the third valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the first valid attempt of the stepping manoeuvre in the Control Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the second valid attempt of the stepping manoeuvre in the Control Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the third valid attempt of the stepping manoeuvre in the Control Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the first valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the second valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the third valid attempt of the stepping manoeuvre in the Intervention Proximal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the first valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the second valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.
Lower limb kinematics - Peak of Rearfoot Eversion | The Lower limb kinematics - Peak of Rearfoot Eversion will be assessed during the third valid attempt of the stepping manoeuvre in the Intervention Distal Condition
  For the capture and analysis of kinematic data during the execution of the stepping manoeuvre, the Vicon movement capture and analysis system will be used.

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

REFERENCES:
- [Derived] Souto LR, Serrao PRMDS, Pisani GK, Tessarin BM, da Silva HF, Machado EM, de Oliveira Sato T, Serrao FV. Immediate effects of hip strap and foot orthoses on self-reported measures and lower limb kinematics during functional tasks in individuals with patellofemoral osteoarthritis: protocol for a randomised crossover clinical trial. Trials. 2022 Sep 5;23(1):746. doi: 10.1186/s13063-022-06676-0. PMID 36064729